CLINICAL TRIAL: NCT00022490
Title: A Phase II Study To Determine The Anti-Leukemic Effects Of STI571 In Combination With Ara-C In Patients With Chronic Myelogenous Leukemia In Chronic Phase
Brief Title: Imatinib Mesylate Plus Cytarabine in Treating Patients With Chronic Myelogenous Leukemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000068822; OHSU-NCI-4653; OHSU-1184 (Other: OHSU IRB); OHSU-HEM-01017-LX (Other: OHSU Knight Cancer Institute); NCI-4653
Record Dates: First submitted 2001-08-10; First posted 2003-01-27 (Estimated); Results first posted 2012-07-11 (Estimated); Last update posted 2016-01-07 (Estimated); Status verified 2015-12

CONDITIONS: Leukemia
Keywords: chronic phase chronic myelogenous leukemia; Philadelphia chromosome positive chronic myelogenous leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Cytarabine; Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cytarabine/ Imatinib Mesylate (Experimental)
  Interventions: Drug: cytarabine; Drug: imatinib mesylate

INTERVENTIONS:
Drug: cytarabine — Once daily subcutaneous injection of Ara-C (Cytarabine) at a dose of 20 mg (10 mg or 5 mg if they have been dose reduced) per square meter of calculated body surface area, on days 15-28 of each sequential 28 day cycle
Drug: imatinib mesylate — Once daily oral administration of STI571 (Imatinib Mesylate) at a dose of 400 mg for 12 months.

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Imatinib mesylate may stop the growth of cancer cells by blocking the enzymes necessary for cancer cell growth.

PURPOSE: This phase II trial is studying giving imatinib mesylate together with cytarabine to see how well it works in treating patients with chronic phase chronic myelogenous leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the rate and duration of complete or major and minor cytogenetic responses after 6 and 12 months of treatment in patients with chronic phase chronic myelogenous leukemia treated with imatinib mesylate and cytarabine.
* Determine the rate and duration of complete hematologic responses after 6 and 12 months of treatment in patients treated with this regimen.
* Determine the rate of molecular response in patients with a complete cytogenetic response after 6 and 12 months of treatment with this regimen.
* Determine the pharmacokinetics of this regimen in these patients.
* Determine the safety of this regimen in these patients.

OUTLINE: This is a nonrandomized, open-label, multicenter study.

Patients receive oral imatinib mesylate on days 1-28 and cytarabine subcutaneously on days 15-28. Courses repeat every 28 days for 12 months in the absence of disease progression or unacceptable toxicity.

Patients are followed for 30-60 days.

PROJECTED ACCRUAL: A total of 15 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Cytogenetically confirmed chronic phase chronic myelogenous leukemia (CML)

  * Less than 15% blasts in peripheral blood or bone marrow
  * Less than 30% blasts and promyelocytes in peripheral blood or bone marrow
  * Less than 20% basophils in blood or bone marrow
  * Platelet count at least 100,000/mm^3
* Philadelphia chromosome positive
* No more than 6 months since initial diagnosis
* No presence of leukemia beyond the bone marrow, blood, liver, or spleen (i.e., chloroma)
* Refused allogeneic stem cell transplantation as first-line therapy

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Eastern Cooperative Oncology Group (ECOG) 0-2

Life expectancy:

* Not specified

Hematopoietic:

* See Disease Characteristics

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* AST or ALT no greater than 2 times ULN

Renal:

* Creatinine no greater than 1.5 times ULN

Cardiovascular:

* No New York Heart Association class III or IV heart disease

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception during and for at least 3 months after study participation
* No other serious uncontrolled medical condition
* No history of noncompliance to medical regimens or potential unreliability

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Disease Characteristics
* No prior biologic therapy for CML

Chemotherapy:

* No prior chemotherapy for CML except hydroxyurea
* Concurrent hydroxyurea to control blood counts during first 3 months of treatment allowed
* No other concurrent chemotherapy

Endocrine therapy:

* No prior endocrine therapy for CML

Radiotherapy:

* No prior radiotherapy for CML

Surgery:

* Not specified

Other:

* More than 28 days since prior investigational anticancer agents
* Prior anagrelide hydrochloride for CML allowed
* Concurrent anagrelide hydrochloride to control blood counts during first 3 months of treatment allowed
* No concurrent grapefruit juice or grapefruit

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2001-06; Primary Completion 2011-05 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian J. Druker, MD, Study Chair — OHSU Knight Cancer Institute
Locations (2):
- United States (2):
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - OHSU Knight Cancer Institute, Portland, Oregon

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cytarabine/ Imatinib Mesylate
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cytarabine/ Imatinib Mesylate
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 21
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 14
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: The Rate of Major Cytogenetic Response at 6 Months
Description: Cytogenetic response is defined in terms of the percentage of Philadelphia (Ph) chromosome. Major cytogenetic response is defined as 0-34% Ph-positive cells.
Time Frame: 6 months
Measure: Number; unit: Participants
Arm/Group | Cytarabine/ Imatinib Mesylate
Number analyzed (Participants) | 24
Participants | 5

2. Secondary Outcome: The Rate of Complete Cytogenetic Response at 6 Months
Time Frame: 6 months
Reporting Status: Not Posted

3. Secondary Outcome: The Rate of Complete and Major Cytogenetic Responses at 12 Months
Time Frame: 12 months
Reporting Status: Not Posted

4. Secondary Outcome: The Rate of Minor Cytogenetic Responses at 6 and 12 Months
Time Frame: 6 and 12 months
Reporting Status: Not Posted

5. Secondary Outcome: The Rate of Complete Hematologic Responses at 6 and 12 Months
Time Frame: 6 and 12 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Cytarabine/ Imatinib Mesylate
Serious Adverse Events (participants affected / at risk) | 13/24
Other Adverse Events (participants affected / at risk) | 0/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cytarabine/ Imatinib Mesylate (N=24)
Neutropenia (Blood and lymphatic system disorders) | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 4
Hyperbilirubinemia (Skin and subcutaneous tissue disorders) | 2
Bone Pain (Musculoskeletal and connective tissue disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 1

LIMITATIONS AND CAVEATS:
Study was terminated, therefore the 12 month response data was not analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes